CLINICAL TRIAL: NCT04295941
Title: Long-term Treatment With Trazodone Once-a-Day (TzOAD) in Patients With MDD: an Observational, Prospective Study
Brief Title: Long-term Study With Trazodone Once-a-Day
Status: Completed | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Responsible Party: Sponsor
Other Study IDs: 039(C)WO19201
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder
Keywords: Trazodone once-a-day; Major Depressive Disorder; Long term therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Trazodone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trazodone once-a-day treated patients: Major Depressive Disorder outpatients who, following an initial positive response to the acute treatment with Trazodone once-a-day monotherapy, will be eligible to enter the continuation therapy and will be observed up to 24 weeks.
  Interventions: Drug: TraZODone Hydrochloride 300 MG

INTERVENTIONS:
Drug: TraZODone Hydrochloride 300 MG — Oral administration of Trazodone once-a-day.

SUMMARY:
The aim of the present observational study is to assess the clinical response, functional impairment and quality of life in outpatients with Major Depressive Disorder who demonstrated an initial positive response to the acute treatment with Trazodone once-a-day monotherapy, for up to 24 weeks.

DETAILED DESCRIPTION:
This is an observational, prospective, single group, multicentre, international study.

The present study is planned to assess, in a real-world setting, the long-term clinical response, functional impairment and quality of life in outpatients with Major Depressive Disorder who, according to the physician's judgment, have responded to the acute monotherapy (6 to 8 weeks of treatment) with Trazodone once-a-day and are eligible to continue Trazodone once-a-day monotherapy according to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients of any ethnic origin ≥18 years old at Baseline. Outpatients who meet the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 or the International Classification of Diseases (ICD)-10 criteria for MDD as their primary diagnosis and presenting with an episode of MDD.

Patients judged as responders to the acute monotherapy with TzOAD after a minimum of 6 and a maximum of 8 weeks of treatment and who are eligible to continue the assigned monotherapy according to the physician's judgement.

Patients legally capable of giving their written consent for participation in the study and for personal data processing and willing to comply with all study procedures.

Exclusion Criteria:

Patients that meet any of the contraindications to the administration of TzOAD according to the approved SmPC.

Patients with previous or current diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, dysthymic or adjustment disorders, mental retardation, organic mental disorders or mental disorders due to a general medical condition.

Patients with previous or current history of a clinically significant neurological disorder, or any neurodegenerative diseases that might compromise the participation in the study.

Patients who are, according to the physician's judgement, at serious risk of suicide.

Patients with substance abuse or dependence (except nicotine dependence), as defined by DSM-5.

Patients participating in any pharmacological or non-pharmacological interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients presenting with Major Depressive Disorder who, following an initial positive response to the acute treatment with Trazodone once-a-day monotherapy, will be eligible according to the physician's judgement, to enter the continuation therapy and will be observed up to 24 weeks.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-improvement scale responders percentage | 24(+4) weeks
  The clinical response expressed as CGI-I responders' percentage at 24 (+ 4) weeks.

SECONDARY OUTCOMES:
Clinical Global Impression-improvement scale responders percentage | 12 (+ 3) weeks.
  The clinical response expressed as CGI-I responders' percentage at 12 (+ 3) weeks.
Clinical Global Impression-improvement scale responders percentage | 18 (+ 3) weeks
  The clinical response expressed as CGI-I responders' percentage at 18 (+ 3) weeks.
Sheehan Disability Scale score | 24-week period
  The functional impairment evaluated over the 24-week period
EQ-5D-5L Quality of life scale | 24-week period
  The quality of life evaluated over the 24-week period

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center Hera EOOD - Clinic/Outpatient Facility, Sofia, Bulgaria